CLINICAL TRIAL: NCT06766292
Title: Clinical, Radiographic and Histologic Assessment of the Osteogenic Potential of Schneiderian Membrane After Maxillary Sinus Lifting: A Randomized Controlled Clinical Trial.
Brief Title: Osteogenic Potential of Schneiderian Membrane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: rehab soliman (Other)
Responsible Party: Sponsor-Investigator, rehab soliman, lecturer of oral and maxillofacial surgery, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 672/2023
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Bone Healing; Sinus Membrane Osteoginicity
Keywords: sinus lifting; maxillary sinus augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): in this group, the patients underwent open sinus lifting surgery and augmentation of the sinuses by xenograft without any additives
  Interventions: Procedure: open sinus lifting with xenograft only
- study group (Experimental): In the study group: 2.0 mm screws were fixed to the lateral wall of the sinus above the superior osteotomy and placed buccopalatally where the schneiderian membrane was elevated and maintained.
  Interventions: Procedure: primary intervention

INTERVENTIONS:
Procedure: primary intervention — In the study group: 2.0 mm screws were fixed to the lateral wall of the sinus above the superior osteotomy and placed buccopalatally where the schneiderian membrane was elevated and maintained. this technique will suspends the membrane in position to allow the blood clot to organized and formation of bone.
  Arms: study group
Procedure: open sinus lifting with xenograft only — ll Patients in this group underwent open sinus procedures to lift the sinus membrane followed by application of the xenograft as an augmentation material xenograft is used instead of autogenous bone graft to avoid the morbidity of the donor side
  Arms: Control Group

SUMMARY:
Maxillary sinus augmentation is commonly performed by creating a space below the Schneiderian membrane which is further filled using autografts, bone graft substitutes, or a combination of both to allow for new bone formation. Recently, a new method called non-grafting sinus floor augmentation has been introduced as an alternative approach. This method is based on the idea of elevating the membrane and supporting it through implant insertion or the use of space-maintaining devices like titanium screws or mesh. This study was conducted to evaluate the efficacy of new bone formation after sinus floor elevation using space maintaining resorbable pins without graft material.

DETAILED DESCRIPTION:
A randomized control trial was performed on 14 patients with partially edentulous or free end saddle posterior maxilla. The patients were divided randomly into two groups. Both groups underwent maxillary sinus open lifting procedure and augmentation using xenograft * as group A and in group B the sinus membrane was elevated and stabilized by resorbable pins** to maintain the created space stable and without grafting. The study was a double blind one (participants and out¬come assessors were blinded throughout the study).

All the surgical procedures were carried out un¬der local anesthesia using infraorbital and posterior superior alveolar nerve block with palatal infiltration. Full thickness mucoperiosteal flap was elevated to expose the lateral wall of the maxillary sinus. Then the maxil¬lary sinus floor elevation using the lateral window technique was performed. A bone window was outlined using a no. 8 diamond bur mounted on straight hand piece with copious irrigation (sterile saline solution) with cautious taken to not penetrate the sinus membrane. The process of bone removal was done through the cortical bone to reach the membrane without perforation. Complete osteotomy along the boundary of the osseous window until the Schneiderian mem-brane. The Schneiderian membrane was carefully elevated till the desired height.

xenograft Preparation: (control group/ group A)

Xenograft was mixed with saline followed by the protocol of graft packed and compacted against inferior walls and to the sides of the antrum until the new available volume created was filled. The lateral window was covered by collagen membrane before flap closure. Resorbable pins (test group/ group B):

In the study group: 2.0 mm screws were fixed to the lateral wall of the sinus above the superior osteotomy and placed buccopalatally where the schneiderian membrane was elevated and maintained. Then the soft tissue flap was readapted and sutured using continuous and interrupted sutures (3-0 resorbable vicryl)

ELIGIBILITY:
Inclusion Criteria:

1. Adult male/female patients above the age of 25.
2. Patients with one or more teeth requiring implant supported dental restoration in atrophic maxilla (unilateral or bilateral).
3. Alveolar bone height less than 4 mm at the defective site.
4. Good oral hygiene.

Exclusion Criteria:

1. Medically compromised patients with conditions contraindicating surgery (eg. uncontrolled diabetics, bisphosphonate intake, radio or chemotherapy).
2. Patients with active infection at or related to the site of surgery (eg. acute sinusitis).
3. Heavy smokers.
4. Patients not indicated for an implant supported restoration at the time of enrollment (eg. active/untreated periodontal disease).

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-08-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
bone height | 8 months
  will be measured using CBCT (Cone Beam Computed Tomography)

SECONDARY OUTCOMES:
histological analysis | 8 months
  will be measured using hematoxylin and eosin stains

CONTACTS AND LOCATIONS:
Overall Officials: rehab soliman, Principal Investigator — Misr International University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No